CLINICAL TRIAL: NCT00915616
Title: The Potential Therapeutic Effect of Melatonin in Gastro-Esophageal Reflux Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Purpose: Treatment
Other Study IDs: Melatonin and reflux
Record Dates: First submitted 2009-06-01; First posted 2009-06-08 (Estimated); Last update posted 2009-06-08 (Estimated); Status verified 2009-06

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Melatonin

ARMS (4):
- control (No Intervention): 9 healthy normal subjects.
- Group II (Active Comparator): Included 9 patients suffering from GERD; receiving melatonin alone for treatment of GERD in a dose of 3 mg once daily at the bed time.
  Interventions: Drug: Melatonin
- Group III, combined group (No Intervention): Included 9 patients suffering from GERD; receiving omeprazole alone for treatment of GERD in a dose of 20 mg twice daily.
- Group IV (Active Comparator): Included 9 patients suffering from GERD receiving omeprazole and melatonin for treatment of GERD in the same dose of each of them.
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin
  Arms: Group II; Group IV

SUMMARY:
Gastro-Esophageal Reflux Disease was defined as a condition that develops when the reflux of stomach contents causes troublesome symptoms and/or complications. Many drugs used for the treatment of GERD such as omeprazole (a proton pump inhibitor) which is widely used anti-ulcer drug and has been demonstrated to protect against esophageal mucosal injury. Melatonin has been found to protect the gastrointestinal mucosa from oxidative damage caused by reactive oxygen species in different experimental ulcer models. The aim of this study is to evaluate the role of exogenous melatonin in the treatment of reflux disease in human either alone and in combination with omeprazole therapy.

ELIGIBILITY:
Inclusion Criteria:

* patient with GERD ranged from 42 to 56 years

Exclusion Criteria:

* patients with cardiac disease
* patients with renal affection
* patients with liver diseases (due to drug induced, autoimmune disease and viral hepatitis)
* patients on the drugs known to affect the GIT motility (phenothiazines, anticholinergics, nitrates or calcium channel blockers) were excluded during the time of conduction of the study or the preceding two weeks

Ages: 42 Years to 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

REFERENCES:
- [Derived] Kandil TS, Mousa AA, El-Gendy AA, Abbas AM. The potential therapeutic effect of melatonin in Gastro-Esophageal Reflux Disease. BMC Gastroenterol. 2010 Jan 18;10:7. doi: 10.1186/1471-230X-10-7. PMID 20082715